CLINICAL TRIAL: NCT06888804
Title: Evaluation of the Effectiveness of Pulsed Radiofrequency Treatment of the Posterior Tibial Nerve in the Management of Chronic Plantar Pain Due to Calcaneal Fracture
Brief Title: Posterior Tibial Nerve PRF for Painful Calcaneal Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTN-RF for calcaneal fracture
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Calcaneus Fracture
Keywords: Pulsed Radiofrequency Treatment; Tibial Nerve
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Tibial Nerve PRF for Painful Calcaneal Fracture (Active Comparator): posterior tibial nerve pulsed radiofrequency for painful calcaneal fracture
  Interventions: Procedure: ultrasound-guided posterior tibial nerve pulsed radiofrequency
- Control (Active Comparator): control group for painful calcaneal fracture
  Interventions: Other: Control Group

INTERVENTIONS:
Procedure: ultrasound-guided posterior tibial nerve pulsed radiofrequency — The posterior tibial nerve (PTN) was identified with a 5-12 MHz linear ultrasonography (US) probe at the level of the medial malleolus, where it runs posterior to the posterior tibial artery. Using the in-plane technique, a 22-gauge, 10-cm radiofrequency cannula was inserted under US guidance and advanced until the tip was adjacent to the nerve. Pulse radiofrequency was applied at 42°C for 240 s with a pulse width of 20 ms.
  Arms: Posterior Tibial Nerve PRF for Painful Calcaneal Fracture
Other: Control Group — No intervention
  Arms: Control

SUMMARY:
Patients who underwent pulsed radiofrequency (PRF) treatment of the posterior tibial nerve under ultrasound guidance, which is routinely performed in our clinic for severe heel pain following a calcaneal fracture, were evaluated through interviews. The assessment was conducted using the Visual Analog Scale (VAS) for pain and the American Orthopaedic Foot and Ankle Society (AOFAS) score.

DETAILED DESCRIPTION:
Pain following a calcaneal fracture can arise from direct injury, traction injury, idiopathic mechanisms such as reflex sympathetic dystrophy/complex regional pain syndrome (CRPS), or nerve damage. Since there is no single standardized definition or diagnosis for post-surgical nerve pain, such cases are described in the literature as neurapraxia, postoperative neuroma, unexplained heel pain, hypersensitive scar, or CRPS. Typically, this type of pain manifests as burning, paresthesia, dysesthesia, and hyperesthesia.

The tibial nerve plays a crucial role in the sensory and motor innervation of the heel. Following a calcaneal fracture, direct nerve injury, compression, or inflammation of the surrounding tissues may contribute to pain. Pulsed radiofrequency (PRF) has been shown to alleviate chronic pain by delivering an electrical field to the nerve tissue at a controlled temperature of <42°C without causing nerve damage. Additionally, there is evidence supporting PRF's effectiveness in pain relief for patients with various chronic conditions.

In our study, the investigators aim to evaluate patients with persistent pain after a calcaneal fracture who have undergone PRF treatment of the posterior tibial nerve. By monitoring these patients immediately after the intervention, we will assess changes in their pain scores. Additionally, the investigators will compare them to patients with post-calcaneal fracture pain who have opted not to undergo the procedure.

ELIGIBILITY:
Inclusion Criteria:

* History of calcaneal fracture
* VAS score >5
* Pain persisting for more than 3 months after the fracture

Exclusion Criteria:

* Presence of other foot pain-causing conditions (e.g., plantar fasciitis, heel spur)
* Additional fractures other than the calcaneus
* Pregnancy
* Coagulopathy or use of antiplatelet medications
* Mental illness impairing decision-making ability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from baseline to 3rd month after treatment
  VAS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
The American Orthopaedic Foot and Ankle Society (AOFAS) | Change from baseline to 3rd month after treatment
  The American Orthopaedic Foot and Ankle Society (AOFAS) score is evaluated under three subcategories: pain, function, and alignment. It includes both objective (function and alignment) and subjective (pain) data. Patients report their pain levels, which are then scored by physicians. Additionally, patients and doctors collaborate to complete the functional and alignment assessments.
  Scores range from 0 to 100, with 100 representing a healthy patient. This scoring system will be assessed pre-procedure, on the day of the procedure, and at the 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)